CLINICAL TRIAL: NCT03580954
Title: Transcranial Magnetic Stimulation in Primary Progressive Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jordi A Matias-Guiu, Principal Investigator. PhD MD, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17/247-E
Record Dates: First submitted 2018-04-17; First posted 2018-07-10 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Primary Progressive Aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive TMS (estimulation) (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- Repetitive TMS (inhibition) (Active Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Stimulation or inhibition using TMS will be delivered guided by a neuronavigator system in different brain regions.

SUMMARY:
Primary progressive aphasia (PPA) is a clinical syndrome characterized by the neurodegeneration of language brain systems. Three main clinical variants are currently recorgnized (nonfluent, semantic, and logopenic PPA). Nowadays, there are no effective treatments for this disorder.

Transcranial Magnetic Stimulation (TMS) is a technique based on the principle of electromagnetic induction of an electric field in the brain. It has been used as a non-invasive therapy in different disorders, such as depression, bipolar disorder, Parkinson's disease, and in the rehabilitation of post-stroke aphasia. Recent studies have shown how repetitive TMS improved language characteristics in Alzheimer's disease, and there are initial data in patients with PPA.

This research project investigates the effect of repetitive TMS in patients with PPA. Investigators will perform a personalized TMS treatment for each patient (brain region, type of stimulation/inhibition, etc.), according to the specific characteristics of each patient and with the final aim to generate a computational model.

ELIGIBILITY:
Inclusion Criteria:

* Must be clinically diagnosed of PPA according to current diagnostic criteria (Gorno-Tempini et al. 2011) with PET-FDG confirmation.
* Clinical Dementia Rating 0-1.

Exclusion Criteria:

* Contraindications for TMS or MRI
* History of epilepsy
* Pregnancy
* Other language disorder previous to the diagnosis of PPA
* Neuroimaging not suggestive of PPA

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in spontaneous speech (main primary endpoint) | 2 months (at baseline and at the end of the treatment)
  Picture and story description task
Changes in oral naming | 2 months
  Object naming test
Changes in reading | 2 months
  Story and words reading test
Changes in repetition | 2 months (at baseline and at the end of the treatment)
  Non-words and sentence repetition task

SECONDARY OUTCOMES:
Changes in brain metabolism | 2 months (at baseline and at the end of the treatment)
  Brain metabolism measured using 18F-FDG-PET
Changes in clinical impression of change | 2 months (at baseline and at the end of the treatment)
  Patient's clinical impression of change (from 0 to 10)
Changes in brain cortical electrical activity | 2 months (at baseline and at the end of the treatment)
  Changes in the brain cortical electrical activity measured using quantitative electroencephalography (EEG)
Changes in global cognition | 2 months (at baseline and at the end of the study)
  Addenbrooke's Cognitive Examination III
Changes in clinical impression of change | 2 months
  Caregiver's clinical impression of change (from 0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos., Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pytel V, Cabrera-Martin MN, Delgado-Alvarez A, Ayala JL, Balugo P, Delgado-Alonso C, Yus M, Carreras MT, Carreras JL, Matias-Guiu J, Matias-Guiu JA. Personalized Repetitive Transcranial Magnetic Stimulation for Primary Progressive Aphasia. J Alzheimers Dis. 2021;84(1):151-167. doi: 10.3233/JAD-210566. PMID 34487043